CLINICAL TRIAL: NCT04450186
Title: Study Pilot - Hybrid EEG/fMRI Neurofeedback in Depressed Patients
Acronym: NEUROFEEDEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC19_9750_NEUROFEEDEP; 2019-A02877-50 (Other: N° ID-RCB)
Record Dates: First submitted 2020-05-12; First posted 2020-06-29 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Depression
Keywords: Neurofeedback
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEG/fMRI neurofeedback (Experimental): Healthy volunteers
  Interventions: Other: EEG/fMRI neurofeedback

INTERVENTIONS:
Other: EEG/fMRI neurofeedback — EEG/fMRI neurofeedback

SUMMARY:
Cognitive impairment is a common residual symptom after a depressive episode and expose patients to a risk of relapsing or therapeutic resistance.

Neurofeedback (using ElectroEncephaloGraphy - EEG or functional Magnetic Resonance Imaging - fMRI) allows patients to self-regulate their cerebral activity, which is supposedly provided through an intelligible and motivating feedback.

Recent results exhibited clinical improvement in depressed patients who underwent a fMRI neurofeedback protocol targeting the amygdala. Furthermore, prefrontal alpha activity was temporally correlated to variations of the BOLD signal in the amygdala. Simultaneous fMRI/EEG neurofeedback is hypothesized to potentialize its antidepressant effect.

Our objective will be to test this assumption by conducting a double-blind randomized trial, and to prove the superiority of bimodal fMRI/EEG neurofeedback over fMRI neurofeedback alone in depressed patients.

An original visual feedback will be provided and validated beforehand by a pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years old
2. Signature of an informed consent after being given clear and loyal oral and written information

Exclusion Criteria:

Related to the volunteer

1. Prior experience of a neurofeedback task

   Related to the MRI
2. Implanted cardiac pacemaker of defibrillator
3. Brain aneurysm clip
4. Cochlear implant
5. Ocular on encephalic metallic foreign body
6. Endoprothesis implanted for less than 4 weeks and ostheosynthesis device implanted for less than 6 weeks.
7. Claustrophobia

   Other criteria
8. Unstable hemodynamic status
9. Acute respiratory failure
10. Alteration of general state or continuous monitoring requirement
11. Other psychiatric condition (DSM-5) such as schizophrenia, substance abuse…
12. Neurological condition or diagnosis of dementia in medical history
13. Undergoing treatment by benzodiazepines or anticonvulsants prescribed less than a month prior to inclusion
14. Undergoing treatment influencing the blood flow prescribed less than three weeks prior to inclusion
15. Protected person (adults legally protected (under judicial protection, guardianship or supervision), person deprived of their liberty, pregnant woman, lactating woman and minor)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
EEG power in alpha band | day 1
  Measurement by an enregistrement in EEG
Cerebral activation in fMRI | day 1
  Measurement by an enregistrement in fMRI

SECONDARY OUTCOMES:
Technology prone behaviour | day 1
  Measurement by Locus of Control Related to Technology (LCRT) (Beier, 2004, French translation Chikhi, 2017) :
  * Description : Subjective 5-point Likert scale. 8 questions. Self-report.
  * Minimal score : 8
  * Maximal score: 40
  * Interpretation : Assessment of the affinity to technology (higher score - better handling). No cut-off.
Anxious personality traits | day 1
  Measurement by State Trait Anxiety Inventory (STAI - Y) (Spielberger, 1983, French translation Spielberger 1993)
  * Description : 4-point Likert scale. 40 questions. Self report.
  * Two parts : State-anxiety (20 questions) and Trait-anxiety (20 questions)
  * Minimal score : 20
  * Maximal score : 80
  * Interpretation : > 65 - very high anxiety, 56-65 - high, 46-55 - average, 36-45 - low, < 35 - very low
Mindfulness skills | day 1
  Measurement by Five Facets Mindfulness Questionnaire (FFMQ) (Baer, 2006, French translation Heeren, 2011)
  * Description : 5-point Likert scale. 39 questions. Self-report. Five facets : Observing, Describing, Acting with awareness, Non-judging of inner experience, Non-reactivity to inner experience
  * Minimal score : 39
  * Maximal score : 195
  * Interpretation : Measure of the tendency to be mindful in daily life (higher score - mindful traits). No cut-off.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Batail, Principal Investigator — CHU Rennes
Locations (1):
- CHU, Rennes, France

IPD SHARING:
Plan to Share IPD: No